CLINICAL TRIAL: NCT02784457
Title: Gonadotropin Releasing Hormone Antagonist in Treatment of Early-onset Severe Ovarian Hyperstimulation Syndrome - a Randomized Controlled Trial
Brief Title: Gonadotropin Releasing Hormone Antagonist in Treatment of Early-onset Severe Ovarian Hyperstimulation Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammed Faris, Lecturer of Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAT-01
Record Dates: First submitted 2016-05-23; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Assisted Reproduction
MeSH Terms: interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GnRHant (Active Comparator): women who received GnRH antagonist
  Interventions: Drug: Cetrorelix
- Control (No Intervention): women who did not receive GnRH antagonist

INTERVENTIONS:
Drug: Cetrorelix
  Arms: GnRHant

SUMMARY:
Efficacy of the use of GnRH antagonist in treatment of those who develop early-onset severe ovarian hyperstimulation syndrome and had cancelled embryo transfer

ELIGIBILITY:
Inclusion Criteria:

* Women who develop early-onset severe ovarian hyperstimulation syndrome after controlled ovarian stimulation using long GnRH agonist protocol and hCG for triggering ovulation.

Exclusion Criteria:

* Women on short or antagonist protocols.
* Women who received GnRH agonist for triggering ovulation.
* Women who had embryo transfer.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of women who needed culdocentesis or paracentesis of the ascitic fluid | within 2 weeks of onset

SECONDARY OUTCOMES:
Number of women who needed hospitalization | within 2 weeks of onset of symptoms
Time to regression of nausea/vomiting | within 2 weeks of onset of symptoms
Time to regression of large ovarian size | within 4 weeks of onset of symptoms

IPD SHARING:
Plan to Share IPD: Undecided